CLINICAL TRIAL: NCT06790212
Title: A Prospective, Randomized Phase II Study Evaluating CAPOX Combined with Ivonescimab (a PD-1/VEGF-A Bispecific Antibody) Versus CAPOX Alone As Neoadjuvant Therapy in Patients with Locally Advanced Colon Cancer.
Brief Title: Neoadjuvant CAPOX Plus Ivonescimab Versus CAPOX for Locally Advanced Colon Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-IIT-0112
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
Keywords: neoadjuvent chemotherapy; CAPOX; AK112; Ivonescimab
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant AK112 combined with chemotherapy (Experimental): Three cycles of neoadjuvant treatment with CAPOX plus Ivonescimab, followed by radical surgery 4 to 5 weeks after the last oxaliplatin dose.
  Interventions: Drug: Ivonescimab; Drug: Oxaliplatin; Drug: Capecitabine
- Neoadjuvant chemotherapy (Active Comparator): Three cycles of neoadjuvant CAPOX treatment, followed by radical surgery 4 to 5 weeks after the last dose of oxaliplatin.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Ivonescimab — 20mg/kg Q3W，D1
  Other Names: AK112
  Arms: Neoadjuvant AK112 combined with chemotherapy
Drug: Oxaliplatin — Oxaliplatin，130mg/m2，D1，Q3W；
Drug: Capecitabine — Capecitabine，1000mg/m2，po，BID，D1-D14，Q3W

SUMMARY:
Neoadjuvant chemotherapy has been validated by several clinical studies to achieve preoperative downstaging and improve survival outcomes in patients with locally advanced colon cancer . Enhancing the efficacy of neoadjuvant treatment further represents a crucial direction for future research.

Recognizing the potential of synergistic effects between immunotherapy and anti-angiogenic therapy, the investigators conducted the present randomized study to explore whether Ivonescimab （a PD-1/VEGF bispecific-antibody）combined with neoadjuvant chemotherapy in locally advanced colon cancer could potentially further improve treatment outcomes.

DETAILED DESCRIPTION:
This phase II, prospective, randomized controlled trial aims to evaluate the efficacy and safety of combining CAPOX chemotherapy with Ivonescimab, a PD-1/VEGF-A bispecific antibody, compared to neoadjuvant CAPOX therapy alone in patients with high-risk recurrent MSS/pMMR-type colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced resectable colon adenocarcinoma (colon cancer located more than 12 cm from the anal verge);
2. Imaging staging is T4, or T3 (with invasion of the muscularis propria ≥5 mm) combined with at least one of the following risk factors: number of metastatic lymph nodes ≥1, extramural vascular invasion (EMVI+), involvement of the mesocolic fascia. (TNM clinical staging (cTNN) according to the 8th edition of AJCC/UICC guidelines);
3. No distant metastasis;
4. At least one measurable lesion ;
5. Immunohistochemical testing of endoscopic biopsy samples by the study center's pathology department confirms diagnosis as pMMR, or genetic testing confirms MSS/MSS-L status (by PCR or NGS method);
6. No prior anti-tumor treatment for colorectal cancer;
7. Age ≥18 years and ≤75 years, regardless of gender;
8. ECOG performance status score 0-1;
9. Signed written informed consent before enrollment;
10. Expected survival of more than 12 weeks;
11. Adequate organ and bone marrow function.

Exclusion Criteria:

1. History of allergic diseases, severe drug allergies, or known allergy to large molecular weight protein formulations or Ivonesimab;
2. Cardiopulmonary insufficiency or hepatic and renal insufficiency that cannot tolerate CAPOX chemotherapy, known allergies to oxaliplatin, capecitabine, irinotecan;
3. Presence of distant metastases;
4. Incomplete or complete bowel obstruction; however, patients can be enrolled if the obstruction is relieved by conservative treatment, intestinal stenting, or colostomy;
5. History of significant bleeding tendency or coagulation disorders;
6. Any of the following complications:

   1. Major gastrointestinal hemorrhage, perforation
   2. Symptomatic cardiac disease (including unstable angina, myocardial infarction, and heart failure)
   3. Uncontrolled diabetes and hypertension
   4. Uncontrolled diarrhea (despite adequate treatment, it still interferes with daily activities)
7. Patients who are using immunosuppressants, systemic, or absorbable topical steroids for immunosuppressive purposes (dose >10 mg/day prednisone or equivalent), and continue to use them within 2 weeks before enrollment;
8. History of uncontrolled cardiac symptoms or diseases;
9. Previous history of thyroid dysfunction that cannot be maintained within normal range despite medication;
10. Use of traditional Chinese medicine immune modulators within 2 weeks before official treatment, or received systemic chemotherapy, immunotherapy, biological therapy, or other anti-tumor treatments including traditional Chinese medicine within 4 weeks prior to enrollment;
11. Previous exposure to immunotherapy, including immune checkpoint inhibitors, immune cell therapy, or any treatment targeting tumor immune mechanisms;
12. Previous exposure to systemic bevacizumab or its biosimilars;
13. Active infection or unexplained fever >38.5°C during screening or before the first dose (patients with fever due to tumor, as determined by the investigator, may be eligible);
14. Objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonia, active tuberculosis, or severely impaired lung function;
15. Congenital or acquired immunodeficiency (such as HIV-infected individuals, HIV 1/2 antibody positive);
16. For patients with positive acute or chronic active hepatitis B, HBV DNA testing must be performed. If the HBV DNA copy number ≤2×10^3 copies/mL or ≤400 IU/mL or below the limit of detection, they may enroll. HBsAg (+) patients should receive antiviral therapy throughout the study period to prevent viral reactivation. For patients who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic antiviral therapy is not required but close monitoring for viral reactivation is necessary;
17. Acute or chronic active hepatitis C (HCV), defined as HCV antibody positive and HCV RNA levels above the limit of detection;
18. Vaccination with live vaccines less than 4 weeks before the start of study medication or likely to occur during the study period;
19. Known history of psychotropic drug abuse, alcoholism, or drug addiction;
20. Pregnant or breastfeeding women, and men and women unwilling to use contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
MPR rate | though 12 weeks neoadjuvant treatment，after surgery completed
  In the primary tumor (PT), ≤10% residual viable tumor (RVT).

SECONDARY OUTCOMES:
Pathologic complete response，pCR | though 12 weeks neoadjuvant treatment，after surgery completed
  Pathological complete response will be made based on assessment of the surgical specimen at the primary treatment site，the absence of any viable tumor cells in the resected primary tumor specimen and all regional lymph node samples.
R0 resection rate | after surgery completed，up to 1 month
  Complete resection of the tumor with negative margins, meaning no residual tumor is present microscopically.
Disease free survival | 2 years
  Defined as the time from randomization to relapse or death, whichever occurred first
Adverse event (AE) | up to 3 years
  The severity of AE and the laboratory findings were graded by the investigators according to Common Terminology Criteria for Adverse Events, version 4. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, MD，phD, Study Chair — Sun Yat-sen University